CLINICAL TRIAL: NCT05040594
Title: Evaluate the Efficacy and Safety of PavéDerm J-Fill Soft Dermal Filler vs. Restylane® Lyft Lidocaine in the Treatment of Moderate to Severe Nasolabial Folds.
Brief Title: Evaluate the Efficacy and Safety of Lidocaine-Containing Hyaluronic Acid Filler in the Treatment of Nasolabial Folds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: YSP-REN3010-001
Record Dates: First submitted 2021-08-22; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Wrinkles Such as Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (right) B (left) (Experimental): Subjects will receive PavéDerm J-Fill Soft Dermal Filler and Restylane® Lyft Lidocaine. One product will be randomized, per NLF.
  Interventions: Device: PavéDerm J-Fill Soft Dermal Filler; Device: Restylane® Lyft Lidocaine
- Treatment B (right) A (left) (Experimental): Subjects will receive Restylane® Lyft Lidocaine and PavéDerm J-Fill Soft Dermal Filler. One product will be randomized, per NLF.
  Interventions: Device: PavéDerm J-Fill Soft Dermal Filler; Device: Restylane® Lyft Lidocaine

INTERVENTIONS:
Device: PavéDerm J-Fill Soft Dermal Filler — Sodium Hyaluronate 20 mg with Lidocaine hydrochloride 3 mg/mL
Device: Restylane® Lyft Lidocaine — Sodium Hyaluronate 20 mg with Lidocaine hydrochloride 3 mg/mL

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PavéDerm J-fill soft dermal filler vs. Restylane® Lyft lidocaine in the treatment of moderate to severe nasolabial folds.

DETAILED DESCRIPTION:
This is a single-center, subject and evaluator blinded, intra-individual, split-face controlled clinical trial. After subjects voluntarily give written consent to the participation in the study, his/her eligibility for the study will be judged through demographic and past & medication history investigation and laboratory test.

Subjects eligible in the screening will be enrolled. Each patient will receive PavéDerm J-Fill Soft Dermal Filler in one nasolabial fold and Restylane Lyft Lidocaine (20 mg/mL Hyaluronic acid with 3 mg/ml Lidocaine hydrochloride) in the other by randomization.

The faces of all subjects are going to be digitally photographed at rest upon every visit. The identical ambient conditions will be used for all photographs and assessments. To ensure blinding status, the subjects will be put on eye mask during injection. On injection day, subjects will receive injections, with at least 60 minute apart, to each nasolabial fold by the treating investigator. The amount of injection will be determined according to the width, length, and depth of the nasolabial folds to ensure optimal correction for each subject. The injected volume will not exceed 1.0 mL in ipsilateral nasolabial fold. The relevant information associated with the injection of the investigational medical device will be documented.

After each injection, the treating investigator will observe subjects through 30 minutes for assessment of adverse events. Subjects will be asked about adverse events at each follow-up visit, and any adverse events will be documented for safety assessment.

Clinical efficacy will be assessed by the appropriately trained evaluator using the WSRS and GAIS under blinded fashion, as well as by subjects using GAIS. Pre-treatment photographs of each subject taken at the pre-treatment (baseline) will be reviewed and will be used for comparison. The blinded evaluator will assess the photographs taken at each visit after the study device administration (photographic assessment). All subjects will perform the self-assessment by comparing their appearance in a mirror against a high-magniﬁcation photograph taken at baseline at each visit after the study device administration. The mirror symmetry will be reminded in all subjects. Under the explanation by the treating investigator or designee, subjects will assess the satisfaction of wrinkle improvement using the GAIS scoring.

Pain is going to be assessed using a patient self-assessment 10-cm visual analogue scale with anchors at 0 m (no pain) and 10 cm (extreme pain).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 20 and 70.
2. Subjects who want to improve bilateral nasolabial folds that are rated as 3 or 4 grades on the WSRS, and same WSRS scores on both sides (both sides are grade 3 or 4 on the WSRS).
3. Subjects with visually symmetrical bilateral nasolabial folds.
4. Subjects who are capable of understanding and comply with the study procedures, instructions, and visit schedule.
5. Subjects who voluntarily decide to participate in the entire course of the trial and provide written consent in the Informed Consent Form.

Exclusion Criteria:

1. Subjects who received an anticoagulant, thrombolytic, antiplatelet therapy or other substances are knownto increase coagulation time (e.g., herbal supplements with garlic or ginkgo biloba), or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within 2 weeks prior to screening.

   -Except for low-dose aspirin (100 mg, up to 300 mg/day) or equivalent.
2. Subjects who received/used a prohibited treatment/procedure as following:

   * Treatment procedure (e.g., bioresorbable fillers, laser/light therapies, botulinum toxin A injections, face lift, facial peels, excisional facial surgery, dermal photorejuvenation clinically significant oral or maxillofacial surgery, etc.) that may interfere with the treatment area or evaluation within 6 months prior to screening as determined by the Principal Investigator.
   * Prescription strength topical retinoids or other topical anti-wrinkle or acne therapies that may interfere with the treatment area or evaluation within 2 weeks prior to screeningas determined by the Principal Investigator.
   * Any oral other anti-wrinkle or acne therapies that may interfere with the treatment area or evaluation within 4 weeks prior to screening as determined by the Principal Investigator.
3. Subjects who received high dose vitamin E (e.g., 400 IU), corticosteroids, or interferon that may interfere with the treatment area or evaluation within 4 weeks prior to screening.
4. The subject who received soft tissue augmentation as following at the investigational medical device injection site within a certain time frame prior to screening:

   -Previous 6 months with bovine collagen; previous 12 months with porcine or human collagen; previous 18 months with hyaluronic acid or hydroxyapatite.
5. The subject who received soft tissue augmentation near the injection site with any of the following at any time:

   -Autologous fat, polymethylmethacrylate or other acrylates, polyacrylamide, polyethylene oxide, polylactic acid, permanent expander prosthesis (e.g., soft-form or silicon), or other implant materials.
6. Subjects with a scar or skin lesion at the investigational medical device injection site that may interfere with the judgment of the treatment effect.
7. Subjects with a history of anaphylaxis or history or presence of multiple severe allergies, allergy to lidocaine or other amide-type anesthetics, hyaluronic acid products, or any component of devices.
8. The subject is, in the Investigator's opinion, at an undue risk based on the precautions, warnings, and contraindications for local lidocaine anesthetics.
9. Subjects with a history of a hypertrophic scar, keloid, or clinically significant skin pigmentation disorders.
10. Subjects with a skin disease or wound infection at the investigational medical device injection site.
11. Subjects who participated in another clinical trial within 60 days prior to screening or plan to participate in another investigation during the course of this study.
12. Pregnant or breastfeeding women or women of childbearing potential who have a plan to get pregnant during the study period, or are not using medically acceptable contraception or not consenting to practice birth control from screening until 30 days after the study has ended (last study procedure).

    * Medically acceptable methods of contraception: non-hormonal intrauterine device or double barrier method (e.g., condom with foam or vaginal spermicidal suppository, diaphragm with spermicide). Complete abstinence can be used as a method of contraception.
    * Be surgically sterile for at least 6 months and/or Post-menopausal for at least 1 year are not considered as women with childbearing potential.
13. History of autoimmune diseases/connective tissue disease, or currently suffer from autoimmune disease/connective tissue disease (e.g., rheumatoid arthritis, Crohn's disease, systemic lupus erythematosus, polymyositis (PM), dermatomyositis (DM) or scleroderma.)
14. Subjects with poorly controlled diabetes mellitus (e.g., an uninterrupted HbA1c >8.0% for ≥1 year despite standard care, are at high risk for complications; standard care with three oral glucose-lowering medications).
15. Subjects with epilepsy, which is not controlled by anti-epilepsy therapy.
16. Subjects with underlying porphyria.
17. Subjects with underlying bleeding disorders.
18. History of malignancy within the past 5 years.
19. Subjects who plan to receive other wrinkle improvement treatment in the lower face (below the lower orbital rim) during this trial.
20. Subjects with underlying systematic diseases (e.g., cardiovascular, digestive, respiratory, endocrine, central nervous system disorders that seems clinically significant), active skin disease or inflammation on or near nasolabial folds that, in the Principal Investigator's opinion, may interfere with treatment area and/or study assessments.
21. Subjects who are otherwise determined by the investigator as ineligible for this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
The Mean change of the Wrinkle Severity Rating Scale scored by the blinded evaluator. | From baseline to Week 24.
  Mean change of the Wrinkle Severity Rating Scale (WSRS) from baseline to Week 24 will be assessed by a blinded evaluator who will judge the severity score from taken photos based on the deﬁnition of WSRS Grades.

SECONDARY OUTCOMES:
The Mean change of the Wrinkle Severity Rating Scale assessed by the blinded evaluator. | From baseline to Week 4 and 12.
  Mean change of the Wrinkle Severity Rating Scale (WSRS) from baseline to Week 4 and Week 12 will be assessed by a blinded evaluator who will judge the severity score from taken photos based on the deﬁnition of WSRS Grades.
Injection pain evaluated by the subjects after injection | 0, and 15, 30, 45, and 60 minutes after the injection.
  Visual Analogue Scale for injection site pain assessment will be evaluated by the subject with anchors at 0 cm (no pain) and 10 cm (extreme pain) after the injection.
The Global Aesthetic Improvement Scale assessed by the blinded evaluator and subjects | At Week 4, 12, and 24
  1. Proportion of subjects with a ≥ 1 point on Global Aesthetic Improvement Scale (GAIS) from baseline to Week 4, 12, and 24 after injection will be evaluated by a blinded evaluator who will judge the severity score from taken photos based on the deﬁnition of GAIS Grades.
  2. Proportion of subjects with a ≥ 1 point on GAIS from baseline to Week 4, 12, and 24 after injection will be evaluated by the subjects based on a live assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chih-Chiang, Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan